CLINICAL TRIAL: NCT02254291
Title: Safety and Efficacy of Semaglutide Once Weekly Versus Sitagliptin Once Daily, Both as Monotherapy in Japanese Subjects With Type 2 Diabetes
Brief Title: A Trial Comparing the Safety and Efficacy of Semaglutide Once Weekly Versus Sitagliptin Once Daily in Japanese Subjects With Type 2 Diabetes
Acronym: SUSTAIN™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9535-4092; U1111-1140-5334 (Other: WHO); JapicCTI-142663 (Registry Identifier: JAPIC)
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Results first posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2017-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Semaglutide 0.5 mg (Experimental)
  Interventions: Drug: semaglutide
- Semaglutide 1.0 mg (Experimental)
  Interventions: Drug: semaglutide
- Sitagliptin 100 mg (Active Comparator)
  Interventions: Drug: sitagliptin

INTERVENTIONS:
Drug: semaglutide — Once weekly doses of 0.5 mg semaglutide after an initial dose escalation step of 0.25 mg (4 weeks). Total duration of treatment is 30 weeks. Administered subcutaneously (s.c. under the skin).
  Arms: Semaglutide 0.5 mg
Drug: semaglutide — Once weekly doses of 1.0 mg semaglutide after an initial dose escalation step of 0.25 mg (4 weeks) followed by 0.5 mg for 4 weeks. Total duration of treatment is 30 weeks. Administered subcutaneously (s.c. under the skin).
  Arms: Semaglutide 1.0 mg
Drug: sitagliptin — Daily doses of 100 mg sitagliptin. Total duration of treatment is 30 weeks. Administered as oral tablets.
  Arms: Sitagliptin 100 mg

SUMMARY:
This trial is conducted in Japan. The purpose is to compare the safety of once-weekly dosing of semaglutide (0.5 and 1.0 mg) versus sitagliptin (100 mg) once daily, both as monotherapy during 30 weeks of treatment in Japanese subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 20 years or older at the time of signing informed consent
* Glycated hemoglobin (HbA1c) between 6.5% and 9.5% (48-80 mmol/mol) (both inclusive) for subjects treated with oral antidiabetic drug (OAD) monotherapy and between 7.0% and 10.5% (53-91 mmol/mol) (both inclusive) for subjects treated with diet and exercise therapy at screening
* Japanese subjects diagnosed with type 2 diabetes who are: a) on stable OAD monotherapy at a half-maximum dose or below according to the approved Japanese labelling in addition to diet and exercise therapy for at least 30 days prior to screening (week -8) (For metformin only: the maximum dose of 750 mg/day is allowed except for METGLUCO®. For METGLUCO®, the allowable half-max dose of 1125 mg/day must be applied.). 'Stable' is defined as unchanged medication and unchanged dose, or b) on stable diet and exercise therapy for at least 30 days prior to screening (week -2)

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method (e.g. abstinence, diaphragm, condom [by the partner], intrauterine device, sponge, spermicide or oral contraceptives) throughout the trial including the 5-week follow-up period
* Treatment with once-weekly glucagon-like peptide-1 (GLP-1) receptor agonists within 90 days prior to screening
* Treatment with any glucose lowering agent(s) (except for pre-trial OAD for subject treated with OAD monotherapy) in a period of 60 days prior to screening. An exception is short-term treatment (7 days or less in total) with insulin in connection with inter-current illness
* Any disorder which, in the opinion of the investigator, might jeopardise subject's safety or compliance with the protocol
* History of chronic or idiopathic acute pancreatitis
* Screening calcitonin value of 50 ng/L (pg/mL) or greater
* Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN2)
* Impaired renal function defined as estimated glomerular filtration rate (eGFR) less than 60 ml/min/1.73 m^2 per modification of diet in renal disease (MDRD) formula (4 variable version)
* Acute coronary or cerebrovascular event within 90 days before randomisation
* Heart failure, New York Heart Association (NYHA) class IV

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2014-10-02 (Actual); Primary Completion 2015-11-11 (Actual); Study Completion 2015-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry GCR, 1452, Study Director — Novo Nordisk A/S
Locations (22):
- Japan (22):
  - Novo Nordisk Investigational Site, Asahikawa-shi, Hokkaido
  - Novo Nordisk Investigational Site, Chitose, Hokkaido
  - Novo Nordisk Investigational Site, Chuo-ku Tokyo
  - Novo Nordisk Investigational Site, Chuo-ku, Tokyo
  - Novo Nordisk Investigational Site, Ebina-shi
  - Novo Nordisk Investigational Site, Izumisano
  - Novo Nordisk Investigational Site, Kashiwara-shi, Osaka
  - Novo Nordisk Investigational Site, Katsushika-ku, Tokyo
  - Novo Nordisk Investigational Site, Kumamoto-shi,Kumamoto
  - Novo Nordisk Investigational Site, Naka-shi, Ibaraki
  - Novo Nordisk Investigational Site, Nishinomiya-shi, Hygo
  - Novo Nordisk Investigational Site, Osaka-shi, Osaka
  - Novo Nordisk Investigational Site, Ota-ku, Tokyo
  - Novo Nordisk Investigational Site, Ōita
  - Novo Nordisk Investigational Site, Sapporo-shi, Hokkaido
  - Novo Nordisk Investigational Site, Shimotsuke-shi, Tochigi
  - Novo Nordisk Investigational Site, Shinjuku-ku, Tokyo
  - Novo Nordisk Investigational Site, Suita-shi, Osaka
  - Novo Nordisk Investigational Site, Takatsuki-shi, Osaka
  - Novo Nordisk Investigational Site, Tokyo
  - Novo Nordisk Investigational Site, Yokohama
  - Novo Nordisk Investigational Site, Yokohama, Kanagawa

REFERENCES:
- [Result] Seino Y, Terauchi Y, Osonoi T, Yabe D, Abe N, Nishida T, Zacho J, Kaneko S. Safety and efficacy of semaglutide once weekly vs sitagliptin once daily, both as monotherapy in Japanese people with type 2 diabetes. Diabetes Obes Metab. 2018 Feb;20(2):378-388. doi: 10.1111/dom.13082. Epub 2017 Oct 5. PMID 28786547
- [Derived] Husain M, Bain SC, Holst AG, Mark T, Rasmussen S, Lingvay I. Effects of semaglutide on risk of cardiovascular events across a continuum of cardiovascular risk: combined post hoc analysis of the SUSTAIN and PIONEER trials. Cardiovasc Diabetol. 2020 Sep 30;19(1):156. doi: 10.1186/s12933-020-01106-4. PMID 32998732
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 25 sites in Japan. These sites randomised/assigned subjects to treatment.
Pre-assignment Details: Subjects were either on stable diet and exercise therapy only or on stable oral anti-diabetic drug (OAD) monotherapy (a maximum dose of 750 mg metformin or 2250 mg METGLUCO according to approved Japanese labelling) in addition to stable diet and exercise therapy for at least 30 days prior to screening (week -8 or week -2).
Groups:
- Semaglutide 0.5 mg: Subjects were randomized to receive semaglutide 0.5 mg once weekly subcutaneously (s.c.; under the skin) in the thigh, abdomen, or upper arm for a duration of 30 weeks. Subjects followed a fixed dose escalation pattern to improve tolerability concerns, starting with once-weekly doses of 0.25 mg for 4 weeks (4 doses), then escalated to 0.5 mg once weekly maintenance dose for 26 weeks (maximum dose). Doses were not changed during the trial after the maintenance dose was reached. Semaglutide 1.34 mg/mL was supplied in a 1.5 mL pre-filled PDS290 pen-injector and administered on the same day of every week during the trial. For subjects previously treated with OAD monotherapy, their 8-week pre-trial OAD was washed out before randomisation. All subjects continued their pre-trial treatment of diet and exercise therapy throughout the trial.
- Semaglutide 1.0 mg: Subjects were randomized to receive semaglutide 1.0 mg once weekly subcutaneously (s.c.; under the skin) in the thigh, abdomen, or upper arm for a duration of 30 weeks. Subjects followed a fixed dose escalation pattern to improve tolerability concerns, starting with once-weekly doses of 0.25 mg for 4 weeks (4 doses), then escalated to 0.5 mg once weekly for 4 weeks, and finally escalated to 1.0 mg once weekly maintenance dose for 22 weeks (maximum dose). Doses were not changed during the trial after the maintenance dose was reached. Semaglutide 1.34 mg/mL was supplied in a 1.5 mL pre-filled PDS290 pen-injector and administered on the same day of every week during the trial. For subjects previously treated with OAD monotherapy, their 8-week pre-trial OAD was washed out before randomisation. All subjects continued their pre-trial treatment of diet and exercise therapy throughout the trial.
- Sitagliptin: The subjects in this arm received oral fixed dose of sitagliptin 100 mg tablet once daily for a duration of 30 weeks. For subjects previously treated with OAD monotherapy, their pre-trial OAD was washed out before randomisation. Doses of sitagliptin were not changed throughout the trial. All subjects continued their pre-trial treatment of diet and exercise therapy throughout the trial.
Period: Overall Study
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Started | 103 | 102 | 103
Exposed | 103 | 102 | 103
Completed | 103 | 99 | 101
Not Completed | 0 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 3 | 1
Not completed — Missing follow-up information | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomised subjects who have received at least one dose of trial product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin | Total
Number analyzed (Participants) | 103 | 102 | 103 | 308
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (10.4) | 58.1 (11.6) | 57.9 (10.1) | 58.3 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 27 | 22 | 73
  Male | 79 | 75 | 81 | 235
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.23 (1.02) | 8.01 (0.85) | 8.20 (0.89) | 8.15 (0.93)

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Emergent Adverse Events (TEAEs)
Description: An adverse events (AEs) was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. All AEs mentioned here are treatment emergent adverse events (TEAE) defined as an event that had onset date (or increase in severity) on or after the first day of exposure to randomised treatment (week 0-30 treatment period) and no later than the follow-up visit during the on-treatment observation period (date of last dose + 42 days).
Time Frame: Weeks 0-30
Population: The safety analysis set (SAS) included all subjects receiving at least one dose of trial product and subjects contributed to the evaluation "as treated".
Measure: Number; unit: Number of events
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 103 | 102 | 103
Number of events | 228 | 197 | 186

2. Secondary Outcome: Number of Severe or Blood Glucose (BG) Confirmed Symptomatic Hypoglycaemic Episodes
Description: Severe or blood glucose (BG) confirmed symptomatic hypoglycaemic episodes were defined as episodes that were severe and/or BG confirmed by a plasma glucose value of <56 mg/dL (3.1 mmol/L), with symptoms consistent with hypoglycaemia. Severe hypoglycaemia was an episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. The episodes mentioned here are treatment emergent hypoglycaemic episodes and defined as an event that had onset date (or increase in severity) on or after the first day of exposure to randomised treatment (week 0-30 treatment period) and no later than the follow-up visit during the on-treatment observation period (date of last dose + 42 days).
Time Frame: Weeks 0-30
Population: as for outcome 1
Measure: Number; unit: Number of episodes
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 103 | 102 | 103
Number of episodes | 0 | 1 | 0

3. Secondary Outcome: Change in Glycosylated Haemoglobin A1c (HbA1c)
Description: Mean changes in HbA1c values from baseline after 30 weeks of treatment. Changes in HbA1c were analysed using a mixed model for repeated measurements (MMRM) with treatment and pre-trial treatment at screening as fixed factors and baseline value as covariate. The data were analysed for the "on-treatment without rescue medication" observation period which includes observations noted at or after the date of first dose of randomised treatment and not after the last dose of the trial product (+ a 7-day visit window) or initiation of rescue medication.
Time Frame: Week 0 and week 30
Population: The full analysis set (FAS) included all randomised subjects who have received at least one dose of trial product. All subjects contributed to the statistical model of the data analysis, but not all subjects had a value at week 30.
Measure: Least Squares Mean (Standard Error); unit: Percentage of glycosylated haemoglobin
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Number analyzed (Participants) | 103 | 102 | 103
Percentage of glycosylated haemoglobin | -1.87 (0.07) | -2.18 (0.07) | -0.74 (0.07)

ADVERSE EVENTS:
Time Frame: All AEs presented here are treatment emergent adverse events (TEAE). A TEAE included events that had onset date (or increase in severity) on or after the first day of exposure (week 0) to randomised treatment (week 0-30 treatment period) and no later than the follow-up visit during the on-treatment observation period (date of last dose + 42 days).
Description: The safety analysis set (SAS) included all subjects receiving at least one dose of the trial product and subjects contributed to the evaluation "as treated".
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Sitagliptin
Serious Adverse Events (participants affected / at risk) | 6/103 | 2/102 | 2/103
Other Adverse Events (participants affected / at risk) | 53/103 | 46/102 | 36/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 0.5 mg (N=103) | Semaglutide 1.0 mg (N=102) | Sitagliptin (N=103)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Postrenal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 0.5 mg (N=103) | Semaglutide 1.0 mg (N=102) | Sitagliptin (N=103)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4) | 7 (8) | 0 (0)
Amylase increased (Investigations) | 6 (7) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 15 (16) | 12 (12) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 9 (10) | 8 (8) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 9 (14) | 2 (3)
Lipase increased (Investigations) | 10 (12) | 7 (8) | 4 (5)
Nasopharyngitis (Infections and infestations) | 17 (21) | 18 (22) | 30 (42)
Nausea (Gastrointestinal disorders) | 11 (12) | 13 (22) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"At the end of the trial, one or more scientific publications may be prepared collaboratively by the Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for less than 60 days to protect intellectual property".